CLINICAL TRIAL: NCT01360255
Title: AFP - L3% and DCP as Tumor Markers in Patients With Hepatocellular Carcinoma (HCC) Treated With Transarterial Chemoembolisation (TACE)
Brief Title: AFP- L3% and DCP as Tumor Markers in Patients With Hepatocellular Carcinoma (HCC) Treated With Transarterial Chemoembolisation (TACE)
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Collaborators: Wako Diagnostics (Industry)
Responsible Party: Principal Investigator, Dominik Bettinger, investigator, University Hospital Freiburg
Other Study IDs: HCC2; DRKS00000812 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2011-05-09; First posted 2011-05-25 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2011-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; transarterial chemoembolisation; liver cancer markers: AFP, AFP-L3% and DCP
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — measurement of tumor markers AFP, AFP-L3 and DCP in serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with TACE: Patients treated with transarterial chemoembolisation (TACE) are included in this clinical trial

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the tumors with an increasing incidence worldwide. Often treatment possibilities are limited and only palliative treatment such as a transarterial chemoembolisation (TACE) is possible. Therapeutic response is evaluated three months after TACE by imaging techniques (CT, MRI). In some HCC patients the tumor marker AFP ( alpha-fetoprotein) is elevated, but not all patients show this elevation. In the last years new tumor markers such as AFP-L3 (subfraction of AFP) and des-y-carboxyprothrombin (DCP) have been examined. In this clinical trial the course of these markers are examined after TACE in order to receive hints if the patient will be a therapeutic responder.

Furthermore the investigators are interested in the quality of life after TACE. Patients receive a questionnaire with regard to the quality of life before and 3 months after TACE.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma (HCC) treated with transarterial chemoembolisation are enrolled in this clinical trial. The aim of this trial is to evaluate the usefulness of the liver cancer markers AFP, AFP-L3% (subfraction of AFP) and des-y- carboxyprothrombin (DCP) after TACE therapy. Some authors could have shown that AFP-L3% is rising in small tumor nodules under 2 cm and so the markers which should decrease after TACE can give a hint for the therapeutic response after the intervention. So the important aim of this trial is to improve the early detection of tumor recurrence after TACE.

Furthermore the quality of life measured by the EORTC QLQ C30 before and after TACE is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80
* diagnosis of HCC according the AASLD criteria
* TACE is planned
* resection is impossible

Exclusion Criteria:

* liver tumor of unknown origin
* other liver tumors
* TACE is impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed hepatocellular carcinoma according to the AASLD criteria and who are treated with transarterial chemoembolisation (TACE) are included in this clinical trial. The patients are recruted in our primary care clinic in the department of gastroenterology and hepatology.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11-15 (Actual)

PRIMARY OUTCOMES:
comparison of liver cancer markers AFP, AFP-L3% and DCP before and after TACE | baseline, 1 month and 3 months
  Liver cancer markers AFP, AFP-L3 and DCP are measured before TACE, 1 month and 3 months after TACE in order to evaluate the course of these markers after the intervention

SECONDARY OUTCOMES:
comparison of quality of life before and after TACE | baseline and 3 months
  analysing the quality of life before and after TACE (3 months after TACE) using the EORTC- QLQ- C30.
long-term survival (1-year, 3-year, 5-year) | up to 5 years
progression- free - time | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Spangenberg, Prof. Dr., Principal Investigator — University Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany